CLINICAL TRIAL: NCT02526069
Title: An ACT Based Application for Young People With Type 1 Diabetes
Acronym: ACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No uptake from potential participants
Sponsor: University of Edinburgh (Other)
Responsible Party: Principal Investigator, Estelle Barker, Trainee Clinical Psychologist, University of Edinburgh
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15-SS-0064
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Acceptance and Commitment Therapy

ARMS (1):
- SweetSpot users (Other): Participants will interact with the smartphone application for as long or as little as they wish. They will be asked to complete questionnaires at baseline (pre), 4 weeks (post), and to attend an interview.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — An application based on Acceptance and Commitment Therapy

SUMMARY:
Study Objectives:

This study aims to assess the feasibility and acceptability of an application utilising Acceptance and Commitment Therapy in young people with type 1 diabetes.

Primary Research Questions:

Is an ACT based application feasible and acceptable to young people with type 1 diabetes.

Study Design:

Patients will use the app for four weeks and then be invited to attend an interview discussing the acceptability, usability and feasibility of the app. Clinician's will also be invited to take part in a workshop where they interact with the app and provide feedback.

Consent for will be obtained through the app. Additional consent for the recording of interviews will be obtained in paper format and stored in a secure locked cabinet at Edinburgh University.

Quantitative data will also be collected on well-being, psychological flexibility, and data usage.

Data Collection

Qualitative feedback:

Interviews will be recorded and transcribed using unique identifiers.

Outcome measures and data usage patterns:

Data will be collected on a password protected database which can only be obtained via a password protected and encrypted server from University of Edinburgh.

Data Analysis:

Phase 1:

Framework analysis and interpretive phenomenological analysis will be utilised to create themes from the qualitative feedback.

DETAILED DESCRIPTION:
Study Design:

The diabetes teams will select participants who meet inclusion criterion and the team will provide them with information leaflets. The information sheets will include contact details of the research team should any queries arise and contact details of somebody independent from the study. Parents/guardians of volunteers between 13-16 years old will also be able to access the information leaflet so they are aware of the study that their child has volunteered to participate in. The information leaflets will provide information surrounding consent. The information sheets will include a uniform resource locator (URL) where patients who have been selected by their diabetes teams will volunteer to download the app (SweetSpot) from.

Once the individual downloads the application or provided with an Android device by the University, they will be required to provide contact details for themselves, their GP and diabetes teams. This is so GP's can be made aware of the patients participation and so diabetes teams can be informed if the research team have concerns regarding an individual. Additionally, participants can be informed of any relevant developments throughout the study and this can be the forum to disseminate findings from the study.

All identifiable data will be stored electronically on a secure local server and password protected database. Any data removed from this database will be partially identifiable through a unique identifier (UID) which will link the two data sets. Analysis will be conducted on fully anonymised data.

Participants who have volunteered to take part in the study will have approximately four weeks to use the app and will be requested to attended an interview to provide feedback on the feasibility and user-friendliness of the app. As well as obtaining consent through the app, patients participating in this phase will provide consent to participate in the focus group.

Additionally, clinicians in the field will be aware of workshops for clinicians to interact with the app. This will be due to the chief investigator attending meetings explaining the study. A follow-up email will be disseminated to the teams with an information sheet and clinicians can volunteer to attend a workshop where they can use the app and provide feedback on the acceptability and feasibility of SweetSpot. Consent will be obtained at the workshop from clinicians.

The general format which each individual will follow contains 6 chapters with individual sessions which have been adapted from "ACT for diabetes self-management" manual. These include:

Chapter 1- Identifying problems.

* Information, consent demographics & baseline questionnaires.
* Barriers to self-management, where barriers direct us.
* Responding to barriers.

Chapter 2 - A choice to be willing.

* Trying something different.
* Letting go of struggles.

Chapter 3-What's important to us.

* Noticing the direction we're moving.
* Choosing our direction.

Chapter 4- How to move towards what we care about.

* Moving towards our values.
* Barriers in moving towards our desired direction.
* Recognising our struggles.

Chapter 5 - How to work flexibly with obstacles.

* School.
* University.
* Work.
* Socialising.
* Family.
* Relationships.

Chapter 6-keeping going.

* How to keep on track.
* Choose what works.

Study Population:

Participants:

The study aims to recruit 12 participants from NHS Lothian, NHS Glasgow & Clyde, NHS Fourth Valley, NHS Dumfries & Galloway, NHS Borders, and NHS Lanarkshire.

Identifying Participants:

Clinician's from diabetes teams in the NHS boards involved will identify patients who meet inclusion criteria and competent to provide consent. These participants will be provided with information leaflets when they attend their regular NHS clinic appointment. A volunteer sample from those selected will pilot SweetSpot. Information leaflets will be available to parents/guardians of patients who are younger than 16 years old. An email address for the chief investigator and a person independent from the research team will also be included in the information leaflet.

Consent Process:

The information sheet containing the URL will state that if they download SweetSpot they are consenting to being involved in an interview to feedback their experience of using SweetSpot which will be recorded and used for research purposes. Participants will be asked to provide their email or phone number so the interview can be arranged, and for future contact should any additional information relevant to the research become available, they will be informed of this and so results can be disseminated via email. The chief investigator will introduce the study to Psychologists in the diabetes network and will visit diabetes teams who have shown an interest in the study to explain it in more detail to the whole team. Further to this an email will be disseminated to NHS diabetes clinicians regarding an educational workshop which introduces SweetSpot, allows clinicians to use SweetSpot and generates feedback from Clinicians regarding acceptability, feasibility and user-friendliness of the app. The workshop will have an information leaflet which will explain that by attending the workshop clinicians are consenting to being involved in a focus group to feedback their experience of using SweetSpot which will be recorded and used for research purposes and a subsequent consent form will be required to be completed at the workshops. It was deemed vital that formative work was conducted in collaboration with targeted users and service providers. Participants will be required to fill in a consent form before the workshops and focus groups. They are required to provide consent for two issues once they volunteer to download the app: 1. to consent to providing contact information of themselves, GP and diabetes team, 2. to consent to their data being used for research purposes. If they do not consent to both these issues they will not be able to access the app content.

There will be direct questions within the app which address consent:

1. Do you consent to your diabetes team being informed of your participation in this study, and that further contact will be made if any concerns about your well-being arise?
2. Do you consent to your data being used for research purposes in this study? If the participant responds no to question 1 or 2, then they will not be able to access the app. The GP and diabetes team will still be informed of their participation in the study. An information leaflet given to potential participants by their health care team will also cover consent issues.

A statement in the information sheets will also state:

By downloading the app you are consent that "I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from the Sponsor (University of Edinburgh), from the NHS organisation or other authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records."

Data Collection:

A unique identifier (UID) is assigned to each participant's data. All data will be stored electronically on an encrypted firewall protected secure local server and password protected database. The measures used to assess effectiveness of the application for self-monitoring behaviours are self-report of blood glucose measurements, insulin injecting, diet and physical exercise imputed daily. The outcome measures will be well-being, diabetes related distress and self-care behaviours.

Data Analysis for Qualitative Data:

The interviews and the workshop will be transcribed and the audio recording will be deleted. Framework analysis will be utilised for the workshop. Interpretive phenomenological analysis will be used for the interviews. This is because these types of analysis lies within the phenomenological school of thought, attempting to understand beliefs and attitudes about a topic. Therefore adopting a realist approach which assumes participants are reporting the truth in their experience. Within the realist framework an inductive approach is adopted to ensure interpretations were grounded in the data. It allows for themes to be generated through the research questions but also from the narratives provided by the participants. Framework analysis aims to report patterns within the data by using a systematic way to interpret information. The method uses a matrix which blends empirical investigation in creative study. Framework analysis has been found useful in analysing focus groups. Themes produced will identify amendments which need to be made for the intervention stage of the study. Interpretive phenomenological analysis is a useful analysis for individual interviews as it generates an in-depth analysis of a person's experience.

Data Analysis for Quantitative Data:

A simple t-test analysis will be conducted if the data is normally distributed, or Wilcoxon-sign if the data is non-normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* 13-22 year olds diagnosed with type 1 diabetes or a clinician working in this field
* Understand English
* Android phone
* If a patient to have been diagnosed for at least 6 months
* Ability to give consent

Exclusion Criteria:

• Young people experiencing significant mental health issues. This includes those who are suicidal, experiencing psychosis, or are severely depressed. This will be assessed by the diabetes team which includes psychologists and those potential participants which meet this exclusion criteria will not be asked to participate in the study by the diabetes or research team.

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility of using SweetSpot | 4 weeks
  Interviews will be conducted

SECONDARY OUTCOMES:
Change in Psychological Flexibility - Diabetes specific (DAAS) | baseline, 4 weeks
  The Diabetes Acceptance and Action Scale (DAAS), is a 42 item measure which measures diabetes acceptance aimed at adolescents with type 1 diabetes (Greco & Hart, 2005). It is scored on a five point likert scale from never true to always true, with approximately half the items being reverse scored. This scale has been revised to form a 14 item version which has been found to have good overall reliability α = 0.796, good reliability for action subscale α =0 .71, and good reliability for avoidance subscale α = 0.78.
Change in Psychological Flexibility (AFQ-Y8) | baseline, 4 weeks
  The Avoidance and Fusion Questionnaire for youths 8 item measure (AFQ-Y8) will be utilised for the generic questionnaire. The AFQ-Y8 (Greco et al., 2008) is an 8 item measure which is measures psychological inflexibility in adolescents. It is scored using a five point likert scale from not at all true to very true. The measure is found to have good reliability α = 0.83.
Change in Diabetes Related Distress (PAID-T) | baseline, 4 weeks
  It has been advised to incorporate the WHO-5 with the Problem Areas in Diabetes (PAID) specific measure (Snoek, 2006). Diabetes related emotional distress will be measured by The Problem Areas in Diabetes-Teen Version (PAID-T). The PAID-T is a 26 item measure scored on a likert scale from one-to-six ascertaining how certain situations have distressed individuals over the past month, showing good reliability α = 0.96 (Weissberg-Benchell & Antisdel-Lomaglio, 2011).
Change in Glucose Management | baseline, 4 weeks
  Participants will be asked to input daily glucose measurements. The average will be calculated at the 4 time points to determine whether there has been an improvement in glucose management
Well-being | baseline, 4 weeks
  The well-being 5 item measure

OTHER OUTCOMES:
Change in Valued Living (BEVS) | baseline, 4 weeks
  Values is broken down into 4 domains: work/education, relationships, personal growth/health and leisure. It measures the things people find important in each of these domains and will be measured utilising the Bull's Eye Value Survey (BEVS: Lundgren et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Estelle L Barker, MSc, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom